CLINICAL TRIAL: NCT02982109
Title: Prediction of Postoperative Pain From Individually Assessed Pain Intensity Levels Associated With Venous Cannulation
Brief Title: Pain Evaluation of Venous Cannulation to Predict Postoperative Pain
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anna P Persson, M.D., Lund University
Other Study IDs: REGSKANE-625361
Record Dates: First submitted 2016-11-28; First posted 2016-12-05 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Postop pain level 1: Minor postoperative pain anticipated
- Postop pain level 2: Might experience postoperative pain
- Postop pain level 3: Moderate pain/substantial surgery performed
- Postop pain level 4: Severe postoperative pain expected/major surgery

SUMMARY:
The investigators have recently reported a relationship between pain induced by peripheral venous cannulation and postoperative pain. The purpose of this study is to validate this method of postoperative pain prediction in a larger cohort subjected to different types of surgery.

DETAILED DESCRIPTION:
* The investigators will study all adult (>18 years old) patients going through surgery at the site during a defined period of time. Before induction of anesthesia participants will be asked to assess (in VAS units) the pain intensity associated with peripheral venous cannulation. The maximum level of postoperative pain intensity will be recorded in the post-anesthesia care unit.
* After the endpoint of the study, the patient records will be reviewed, and de-identified relevant data be recorded and analyzed in the Statistical Package for the Social Sciences (SPSS) software.
* Sample size assessment: In a previous study patients scoring ≥ 2.0 on venous cannulation assessed their median pain postoperatively at 5.8 VAS units compared with 2.9 in those scoring < 2.0 - corresponding to a difference in maximum postoperative pain intensity of almost three VAS units. To statistically confirm, with unpaired non-parametric tests, 80 % power (β), and 95% probability (1- α), half of that difference (1.5 VAS units) in pain intensity level between patients scoring above or below 2.0 VAS units, respectively, would require 55 patients in each group subjected to the same kind of surgery. With 4 groups of cases and controls 440 patients would need to be included. As the study is strictly observational, 600 patients will be included to make up for possible missing data.
* Statistics: The Mann-Whitney U- test will be used to compare differences in postoperative pain intensity levels, and the Pearson Chi-square test to compare proportions of patients with moderate or severe postoperative pain, in patients differing in pain scores (above or below 2.0 VAS units) on venous cannulation. Logistic regression analysis will be used to adjust for gender and age and to evaluate the predictive ability of proposed method.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Scheduled for surgery in Halmstad
* Prepared for surgery in the preoperative ward or ward 71 (day-case or direct admittance)

Exclusion Criteria:

* Inability to handle the Visual Analog Scale
* Hospitalized already before surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery at Hallands Hospital Halmstad
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Maximum postoperative pain intensity (0.0-10.0 VAS units) | 2 hours after surgery
  Patients scoring their pain associated with venous cannulation to <2 VAS units will be compared to patients scoring ≥2 VAS units considering median level of maximum postoperative pain intensity.

SECONDARY OUTCOMES:
Risk of developing moderate to severe postoperative pain | 2 hours after surgery
  Proportion of patients with moderate or severe (≥4 VAS units) postoperative pain will be compared between groups of patients scoring </≥ 2 VAS units on peripheral venous cannulation.
Influence of gender | 2 hours after surgery
  With logistic regression analysis investigate the potential influence of gender on the predictive ability of this test.

CONTACTS AND LOCATIONS:
Overall Officials: Anna KM Persson, M.D, Principal Investigator — Lund University
Locations (1):
- Hallands Hospital Halmstad, Halmstad, Halland County, Sweden

IPD SHARING:
Plan to Share IPD: No